CLINICAL TRIAL: NCT07115836
Title: Standard Versus "Single Loop" Bypass After Parietal Gastrectomy: a Randomized Double-blind Study
Brief Title: Standard Versus "Single Loop" Bypass After Parietal Gastrectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Fondation de l'Institut universitaire de cardiologie et pneumologie de Québec (Unknown)
Responsible Party: Principal Investigator, Laurent Biertho, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Second stage SADI, pilot study
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Obesity, Morbid; Obesity
Keywords: Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Intervention Model Description: This is a single-center double-blind randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biliopancreatic diversion with duodenal switch (Active Comparator): Patient randomized for a the standard duodenal switch as second stage surgery after a sleeve gastrectomy (100cm common channel and 150cm alimentary limb)
  Interventions: Procedure: Standard duodenal switch
- Single-anastomosis duodenal-ileal anastomosis (Experimental): Patient randomized for a single-anastomosis duodeno-ileal anastomosis as second stage surgery after a sleeve gastrectomy (250cm common channel)
  Interventions: Procedure: Single-anastomosis duodenal switch

INTERVENTIONS:
Procedure: Standard duodenal switch — Standard duodenal switch as second stage surgery after a sleeve gastrectomy (100cm common channel and 150cm alimentary limb)
  Arms: Biliopancreatic diversion with duodenal switch
Procedure: Single-anastomosis duodenal switch — Single-anastomosis duodeno-ileal anastomosis as second stage surgery after a sleeve gastrectomy (250cm common channel)
  Arms: Single-anastomosis duodenal-ileal anastomosis

SUMMARY:
Bilio-pancreatic bypass (BPD-DS) is the most effective type of bariatric surgery in terms of weight loss and treatment of obesity-related comorbidities such as type 2 diabetes. Nevertheless, the spread of this procedure is limited by the technical difficulties and long-term nutritional complications inherent in this operation.

Recently, a simplified "Duodenal Switch" technique has been proposed. This technique is known as "Single Anastomosis Duodeno-Ileal bypass" (SADI) and involves connecting the duodenum to the ileum, 250 cm upstream of the ileo-caecal valve, via an "omega" loop. This surgery is technically simpler and possibly less risky (particularly from a nutritional point of view) than the "standard" technique developed at the IUCPQ. This explains the enthusiasm in the surgical community for SADI, although the scientific evidence is very limited. The investigator has therefore initiated a prospective randomized study to compare standard bypass with single loop bypass as primary surgery.

In this study, the investigator aims to evaluate the results of SADI versus standard bypass, as 2nd-stage surgery after parietal gastrectomy.

The hypothesis is that SADI will be accompanied by fewer digestive and nutritional side effects, but also by a lower weight loss and a lower rate of recovery from comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a parietal gastrectomy more than 18 months ago and
* Who still meet NIH criteria for bariatric surgery (BMI ≥ 35kg/m2 with associated disease or BMI ≥ 40kg/m2) or
* Have lost < 50% of their excess weight, or
* Have significant weight regain (≥ 20% EWL)
* Accepting long-term care and follow-up and willing to participate in this study after informed consent

Exclusion Criteria:

* Other bariatric procedures apart from parietal gastrectomy.
* Psychiatric illness not stabilized for more than 6 months
* Severe illness with life-threatening consequences within 5 years
* Diagnosis of cancer within the last 3 years
* Chronic digestive disorders (chronic diarrhea, inflammatory diseases, cirrhosis, intestinal resections, functional abdominal pain)
* Pregnancy or desire for pregnancy within 2 years
* Intellectual retardation making consent impossible or patient under guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2028-01-06 (Estimated)

PRIMARY OUTCOMES:
Weight loss | from baseline to 60 months
  % Excess weights loss

SECONDARY OUTCOMES:
Mortality rate | from baseline to 60 months
  Mortality rate
Early complications | from baseline to 30 days
  Complication (≤30 days) graded with Clavien classification
Late complications | from 30 days to 60 months
  Complication (>30 days to 60 months) ga=raded with Clavien classification
Operating time | baseline
  Operating time in minutes
Blood loss | baseline
  Peroperative blood loss (ml) as reported in the operating room
Hospital stay | baseline
  length of hospital stay (days)
Change in quality of life (QLaval) | from baseline to 60 months
  Change in quality of life assessed by the Laval questionnaire evaluating 6 aspects on a scale from 0 to 7, higher scores indicate better quality of life
Change in quality of life (SF36) | from baseline to 60 months
  change in quality of life assessed with the 36-item short form survey evaluating quality of life on a scale form 0 to 100, higher scores indicate better quality of life
Digestive side effects (GERD) | from baseline to 60 months
  Evaluation of gastro-oesophageal reflux symptoms using the GERD Score questionnaire, on a scale from 0 to 72, higher scores indicating greater symptoms
Digestive side effects (LARS) | baseline to 60 months
  Evaluation of bowel function using the LARS questionnaire, on a scale from 0 to 42, with higher scores indicating greater symptoms
Digestive side effect (GIQLI) | from baseline to 60 months
  Evaluation of digestive side effect using the Laval digestive problems evaluation questionnaire, on a scale from 0 to 144, with higher scores indicating less negative impact of symptoms
Malnutrition rate | from baseline to 60 months
  Malnutrition rate using albuminemia (mild 30-34.9g/L; moderate 25-29.9g/L; severe <25g/L)
Nutrient deficiency rate | from baseline to 60 months
  Nutrient deficiency rate based on blood analysis of vitamine A, vitamin D, vitamin B12, Calcium, magnsium, phosphorus, iron, ferritin, TIBC and parathormone and the required dose of supplements
Resolution of associated comorbidities | from baseline to 60 months
  Type 2 diabetes, hypertension, sleep apnea and dislipidemia evolution are evaluated according to treatment, symptoms, vital signs and blood test results to determine whether there has been resolution, improvement, no change, deterioration, or recurrence of the condition according to the criteria of the American Society for Metabolic & Bariatric Surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Criucpq-Ul, Québec, Quebec, Canada